NCT Number: NCT03480282

Official Title: Discussing Stopping Cancer Screening and Prognosis With Older Adults

Document Type: Informed Consent

Document Date: 03/20/2019



\*\*For CCI Use Only\*\*

Approved by the Beth Israel Deaconess Medical Center Committee on Clinical Investigations:

Clinical Investigations:

Consent Approval Date: 03/20/2019

Protocol Number: 2016P000244



## INFORMED CONSENT FORM TO TAKE PART IN A RESEARCH STUDY

Discussing Stopping – Phase 1 - Patients

**SUBJECT'S NAME:** 

TITLE OF RESEARCH PROTOCOL: Discussions of Prognosis and Stopping Cancer Screening in

Older Adults

PRINCIPAL INVESTIGATOR: Mara A. Schonberg, MD, MPH

PROTOCOL NUMBER: 2016-P-000244

#### INTRODUCTION:

- This is a research study;
- Your participation is voluntary;
- > A research study includes only people who choose to take part;
- You may or may not benefit from participating in the study. However, your participation may help others in the future as a result of knowledge gained from the research;
- You may leave the study at any time;
- ➤ If you choose not to take part, or if you leave the study, your decision will in no way harm your relationship with any member of the research team or any other individuals at Beth Israel Deaconess Medical Center

Please read this consent form carefully and ask the investigators or study staff to explain any words or information that you do not clearly understand. Once you read this consent form and understand what your participation in this study will involve, you will be asked to sign this form if you wish to take part. You will be given a signed copy of the form to keep for your records.

# DISCLOSURE OF SPECIAL INTERESTS OF BIDMC AND INVESTIGATORS

This study is being conducted by *Dr. Mara Schonberg* and is funded by the NIH. The funding agency in this study, the NIH, is paying Beth Israel Deaconess Medical Center *and Dr. Schonberg* to perform this research. BIDMC or Dr. Schonberg has *no* additional interests in this research project.

# WHOM TO CONTACT IF YOU HAVE QUESTIONS OR PROBLEMS

If you have any questions, concerns or complaints about this research or experience any problems, you should contact Dr. Mara Schonberg at [617] 754-1414.



TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND

STOPPING CANCER SCREENING IN OLDER ADULTS

PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH

PROTOCOL #: 2016-P-000244



#### **PURPOSE**

The purpose of this study is to learn from patients how they would like their primary care physician (PCP) to talk to them about stopping cancer screening.

## STUDY PARTICIPANTS

You have been asked to be in the study because you are an adult aged 76-89 who undergoes routine cancer screening.

We will conduct focus groups and individual interviews with adults aged 76-89 years, their family members and their PCPs to learn the best language and approach for PCPs to use when talking to older adults about their prognosis and when to stop cancer screening. We will use the data from these focus groups and interviews to develop strategies for PCPs to discuss prognosis with their patients when discussing stopping cancer screening.

Approximately 30 people will take part in this study at Beth Israel Deaconess Medical Center.

## **DESCRIPTION OF STUDY DETAILS**

## 1) Screening

Through medical record review, we will identify adult patients aged 76-89 who undergo routine cancer screening. With permission from you physician, we will contact you about your willingness to participate in the study.

## 2) Study procedures

If you agree to be in this study, you will be asked to read and sign this consent form. After you sign the consent form, the following things will happen:

If you qualify to take part in this research study, a research assistant will ask you some questions about your health and your background. After completing these questions, the research assistant will ask you to participate in an individual interview that will be recorded. As part of the interview, you will be asked whether your doctor has ever talked to you about stopping cancer screening and how you would like your doctor to approach talking to you about stopping cancer screening. The interviewer will also ask you if your doctor has offered to talk to you about your life expectancy and whether you would like your doctor to talk to you about your life expectancy and how you would like your doctor to approach this topic. We will use the information we learn during these interviews to develop strategies for doctors to use when talking to older adults about stopping cancer screening and their life expectancy.

## 3) Monitoring/follow up

This is a one-time study visit. There will be no monitoring or follow up.



TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND

STOPPING CANCER SCREENING IN OLDER ADULTS

PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH




#### RISKS AND DISCOMFORTS

This study poses very little risk to participants. Some participants may develop feelings of anxiety, distress, or fatigue when answering interview questions. You may stop interviews at any time, skip any question that makes you feel uncomfortable, and/or withdraw your participation..

Participant responses and data will be directly and securely stored and password protected via REDCap (web-based software for data collection for research purposes). Interview recordings will be transcribed verbatim through a secure, HIPPA-compliant transcription service. Recordings and transcripts will be stored in a locked cabinet in Dr. Schonberg's office. Each recording will be labeled with a unique study ID and not participant identifiers. Recordings will be heard only for research purposes by the research team and they will be destroyed in compliance with NIH policy. All data for a participant will be linked through their unique study ID. Responses to interview questions will be completely confidential. All interviews will be conducted in private office space or clinical space, or at the patient's home.

## LOSS OF CONFIDENTIALITY

There is the potential for loss of confidentiality by participating in this study. Every effort will be made to protect the confidentiality of your identifiable information.

## CONFIDENTIALITY

Information learned from your participation in this study and from your *medical record* may be reviewed and photocopied by the Food and Drug Administration (FDA) and/or other federal and state regulatory agencies, and by the accreditation agencies, the Committee on Clinical Investigations, the Human Subjects Protection Office and others involved in research administration of the Beth Israel Deaconess Medical Center with protection of confidentiality so far as permitted by applicable law. Information resulting from this study and from your *medical record* may be used for research purposes and may be published; however, you will not be identified by name in such publications.

#### CERTIFICATE OF CONFIDENTIALITY

The National Institutes of Health has issued a Certificate of Confidentiality for this research. This adds special protection for the research information and specimens that may identify you. The researchers may not disclose information or specimens that may identify you, even under a court order or subpoena, unless you give permission. However, a Certificate of Confidentiality does not prevent researchers from disclosing your information or specimens if required by law (such as to report child abuse, communicable diseases or harm to self or others); if you have consented to the disclosure (such as for your medical treatment); or for use in other research as allowed by law. In addition, the Certificate cannot be used to refuse a request if a governmental agency sponsoring the project wants to audit the research. By signing this form, you are giving your consent to the disclosure of your information or specimens for any purpose you have agreed to in this informed document and for any purpose permitted without additional authorization in the BIDMC Notice of



TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND STOPPING CANCER SCREENING IN OLDER ADULTS

PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH




Privacy Practices. Any research information that is placed in your medical record would not be covered under this Certificate. The Certificate does not stop you from voluntarily releasing information about yourself or your involvement in this research. If others obtain your written consent to receive research information or specimens, then the researchers are permitted, but not necessarily required, to disclose that information. **POSSIBLE BENEFITS**It is not possible to predict whether you will benefit directly from participation in this study. However, your participation may help others in the future as a result of knowledge gained from the research.

#### OTHER AVAILABLE OPTIONS

Taking part in this study is voluntary. You have the option to not enroll in the study.

#### IF YOU DECIDE NOT TO TAKE PART IN THE STUDY

Participation in this study is voluntary. You have the right to decide not to take part in this study. If you choose to participate, you have the right to leave the study at any time. Your decision to not participate will not result in any penalties or loss of benefits to you. The investigators will tell you about new information that may affect your willingness to stay in this study.

If you decide not to participate in the study or decide to leave the study early, your decision will not affect your relationship with the research team or any other individual at Beth Israel Deaconess Medical Center.

## INVESTIGATORS RIGHT TO STOP THE STUDY

The investigators have the right to end your participation in this study if they determine that you no longer qualify to take part, or if it would be dangerous for you to continue, or if you do not follow study procedures as directed by the investigators. Beth Israel Deaconess Medical Center or the funding source may stop the study at any time.

## **COSTS AND/OR PAYMENTS TO YOU**

## **COSTS COVERED BY STUDY**

You will not be charged for *anything* that is part of this research study.

#### PAYMENTS TO YOU:

As an appreciation of your time, we will offer \$25 by mailed check for participating in the study.

It may take up to 8 weeks for you to receive payment by check.

Any payments made to you may be taxable income to you. This does not include any payments you may receive to reimburse (pay you back) you for certain expenses like parking fees or travel. We are required to obtain your name and social security number for preparation and submission of Internal Revenue Service (IRS) Form 1099-Misc. You may receive an Internal Revenue Service Form 1099 from BIDMC if you receive more than \$600 or more in one calendar year for taking part

PI Revision Date: 05/23/2018



TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND STOPPING CANCER SCREENING IN OLDER ADULTS

PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH




in one or more research studies at BIDMC. Questions about your own tax status should be referred to your personal tax advisor.

# AUTHORIZATION FOR USE AND DISCLOSURE OF YOUR PROTECTED HEALTH INFORMATION

As part of this study, we will be collecting, using and sharing with others information about you. Please review this section carefully as it contains information about the federal privacy rules and the use and disclosure of your information.

## PROTECTED HEALTH INFORMATION [PHI]

By signing this informed consent document, you are allowing the investigators and other authorized personnel to use [internally at BIDMC] and disclose [to people and organizations outside the BIDMC workforce identified in this consent] health information about you. This may include information about you that already exists (for example: your medical records and other sources of health information, demographic information, the results of any laboratory tests, and mental health records if applicable as well as any new information generated as part of this study. This is your Protected Health Information.

People/Groups at BIDMC Who Will Share and Use Your Protected Health Information may be shared with and used by investigators working on this study, including the supporting research team (such as research assistants and coordinators, statisticians, data managers, laboratory personnel, pharmacy personnel, and administrative assistants), and may also be shared and used by other health care providers at BIDMC who have treated you in the past and have information relevant to the research, or who provide services to you in connection with the research. Your Protected Health Information may also be shared with the members and staff of the Committee on Clinical Investigations of Beth Israel Deaconess Medical Center, which is responsible for reviewing studies for the protection of the research subjects.

# PEOPLE/GROUPS OUTSIDE OF BIDMC WITH WHOM YOUR PROTECTED HEALTH INFORMATION WILL BE SHARED

We will take care to maintain confidentiality and privacy about you and your Protected Health Information. We may share your Protected Health Information with the following groups so that they may carry out their duties related to this study:

- The funding source and/or sponsor of this study, the NIH, and, where applicable, the people and companies that the funding source and/or sponsor use to oversee, administer, or conduct the research (for example, clinical research organizations are companies that are sometimes hired by research sponsors to help manage and run a clinical research study)
- The other hospitals and medical centers taking part in this study and research collaborators at those institutions
- Any external health care providers who provide services to you in connection with this

Informed Consent – Part D CCI Form: 9-2015

PI Revision Date: 05/23/2018



TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND STOPPING CANCER SCREENING IN OLDER ADULTS

PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH




#### research

- Laboratories not affiliated with BIDMC that are involved in conducting tests related to the research
- Statisticians and other data monitors not affiliated with BIDMC
- The members and staff of any other IRBs (beyond the BIDMC Committee on Clinical Investigations) that oversee the research
- Centralized data collectors
- Your health insurance company
- The Food and Drug Administration [FDA], the Department of Health and Human Services [DHHS], the National Institute of Health [NIH], the Office for Human Research Protections [OHRP], and other federal and state agencies that may have jurisdiction over the research
- Hospital and Clinical Research Accrediting Agencies
- Data and Safety Monitoring boards that oversee this study (if applicable)

Those who receive your Protected Health Information during the course of the research may not be required by the federal privacy regulations to protect it, and they may make further disclosures to others and use your information without being subject to penalties under those laws.

## WHY WE ARE USING AND SHARING YOUR PROTECTED HEALTH INFORMATION

The main reason for using and sharing your Protected Health Information is to conduct and oversee the research as described in this Informed Consent Document. There are many other reasons beyond the research for which BIDMC may use or disclose your Protected Health Information. Not all of these reasons require your express written authorization. For example, we will use and share your Protected Health Information to ensure that the research meets legal, institutional and accreditation requirements and to conduct public health activities. The various ways in which BIDMC may use and disclose your protected health information without your authorization are explained in a document called the Notice of Privacy Practices. If you have not received a copy of BIDMC's Notice of Privacy Practices, please ask us for one and review it before signing this form. In addition to signing this document, you may also be asked to sign a BIDMC General Agreement form acknowledging that you have received the BIDMC Notice of Privacy Practices.

## No Expiration Date - Right to Withdraw Authorization

Your authorization for the use and disclosure of your Protected Health Information in this Study shall never expire. However, you may withdraw your authorization for the use and disclosure of your Protected Health Information at any time provided you notify the Principal Investigator in writing. If you would like to take back your authorization so that your Protected Health Information can no longer be used in this study, please send a letter notifying the Principal Investigator of your withdrawal of your authorization to <a href="Dr. Mara A. Schonberg">Dr. Mara A. Schonberg</a> at 330 Brookline Ave., Boston, MA 02215. Please be aware that the investigators in this study will not be required to destroy or retrieve any of your Protected Health Information that has already been used or disclosed before the Principal Investigator receives your letter, and they are permitted to continue to use and disclose



TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND STOPPING CANCER SCREENING IN OLDER ADULTS

PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH




your previously collected information as necessary to complete the research.

## **REFUSAL TO SIGN**

Your clinical treatment may not be conditioned upon whether you sign the Authorization for Research. However, if you choose not to sign this informed consent document and authorization for the use and disclosure of your Protected Health Information, you will not be allowed to take part in the research study.

## RIGHT TO ACCESS AND COPY YOUR PHI

If you wish to review or copy your Protected Health Information as it is made part of your medical record, you may do so after the completion or termination of the study by sending a letter to the Principal Investigator requesting a copy of your Protected Health Information. You may not be allowed to inspect or copy your Protected Health Information until this study is completed or terminated.

#### OTHER IMPORTANT INFORMATION

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a> as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## ADDITIONAL CONTACT FOR QUESTIONS OR CONCERNS

You may contact the Human Subjects Protection Office at [617] 975-8500 in the event that you would like to obtain information or to offer input about the research study. This office is independent of the investigator or investigator's research staff and can also assist with questions relating to your rights as a participant in research, which may include questions, concerns or complaints about your participation in the study.



| SUBJECT'S NAME: |
|---|
| TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND STOPPING CANCER SCREENING IN OLDER ADULTS |
| PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH |



# THE FOLLOWING PARAGRAPHS CONTAIN SOME STANDARD INFORMATION WHICH GENERALLY APPLIES TO INDIVIDUALS PARTICIPATING IN A RESEARCH STUDY.

## CONSENT FORM FOR CLINICAL RESEARCH

I have read the previous page[s] of the consent form and the investigator has explained the details of the study. I understand that I am free to ask additional questions.

If I wish additional information regarding this research and my rights as a research subject, or if I believe I have been harmed by this study, I may contact the Human Subjects Protection Office (HSPO).

I am aware that this is a research project and that unforeseen side effects may occur.

I understand that the Beth Israel Deaconess Medical Center has no formal program for compensating patients for medical injuries arising from this research. Medical treatment will be provided for injuries at the usual charge to me or to my insurer unless payment is otherwise provided for in this consent form.

I understand that participation in this study is voluntary and I may refuse to participate or may discontinue participation at any time without penalty, loss of benefits, or prejudice to the quality of care which I will receive.

I acknowledge that no guarantees have been made to me regarding the results of the treatment involved in

| this study, and I consent to participate in the | study and have been given a | a copy of this form | 1. |
|---|---|---|---|
| Signature of Subject or<br>Legally Authorized Representative<br>(Parent if the subject is a minor) | Date | | |
| Relationship of Legally Authorized Represent | tative to Subject | | |
| The subject has been given the opportunity to h | o read this consent form and as been given a copy. | to ask questions k | efore signing, and |
| SIGNATURE OF INV | VESTIGATOR/Co-Investigator | DATE | _ |
| PRINT INVESTIG | GATOR'S/Co-Investigator's | NAME | - |

A signing co-investigator must be listed on the study's approved Research Staffing Form at the time of consent.

PI Revision Date: 05/23/2018



| SUBJECT'S NAME: |
|---|
| TITLE OF RESEARCH PROTOCOL: DISCUSSIONS OF PROGNOSIS AND STOPPING CANCER SCREENING IN OLDER ADULTS |
| PRINCIPAL INVESTIGATOR'S NAME: MARA A. SCHONBERG, MD, MPH |

APPROVED BY THE

COMMITTEE ON CLINICAL INVESTIGATIONS
03/15/2020

APPROVAL EXPIRATION DATE

# THE FOLLOWING SECTIONS ARE NOT NEEDED FOR ALL STUDIES AND SHOULD BE UTILIZED AS INDICATED:

| If the subject is able to speak and understand English but is not able to read or write |
|---|
| I was present during the entire oral presentation of the informed consent and witnessed the subject's agreement to participate in the study. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: ——— |
| If the subject is able to understand English but is not physically able to read or write or see |
| I was present during the entire oral presentation of the informed consent and witnessed the subject's agreement to participate in the study. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: |
| If the subject is not English speaking and signed the translated Short Form in lieu of the English consent document. |
| As someone who understands both English and the language spoken by the subject, I interpreted, in the subject's language, the researcher's presentation of the English consent form. The subject was given the opportunity to ask questions. |
| Signature of Interpreter: |
| Printed name of Interpreter: |
| Date: |